CLINICAL TRIAL: NCT05711784
Title: A Randomized, Double-blinded, Placebo-controlled, Single-Centre, Comparative, Clinical Safety and Efficacy Study in Subjects With Overweight or Obese Class - I, to Evaluate the Degree of Significant Weight Loss by Regular Intake of Phaseolean (White Kidney Bean Standardized Extract).
Brief Title: A Clinical Safety and Efficacy Study in Subjects With Overweight or Obese Class - I, to Evaluate the Degree of Significant Weight Loss by Regular Intake of Phaseolean (White Kidney Bean Standardized Extract)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NovoBliss Research Pvt Ltd (Other)
Collaborators: Ambe Phytoextracts Pvt. Ltd (Industry)
Responsible Party: Principal Investigator, Dr Nayan Patel, Principal Investigator - Medical Director, NovoBliss Research Pvt Ltd
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NB220038-AG
Record Dates: First submitted 2023-01-13; First posted 2023-02-03 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Body Weight in the Overweight and Obese Class - I Population
MeSH Terms: interventions — Capsules

STUDY DESIGN:
Intervention Model Description: Randomized, Three-arm, Comparative, Double-blinded, Placebo-controlled, Single-center, Dose-response, Safety and Efficacy
Who Masked: Participant, Investigator
Masking Description: Subjects will be randomly assigned in a 1:1:1 ratio to receive either treatment A or B or C. The randomization code will be generated by NovoBliss Research. The randomization schedule will be maintained under controlled access. Double Blind will be followed.
  The Investigator/Evaluator will be blinded to the randomization schedule. The sequence number as per the randomization schedule will be used as Randomization ID.
  Subjects will be randomly allocated to one of the three treatment groups, as per the randomization code. Neither the subject nor the Investigator/Evaluator shall be aware of the treatment allocation (Double Blind). To maintain blinding, the study staff who involves in treatment dispensing and distribution will not be involved in any other study-related activities.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phaseolean (White Kidney Bean Standardized Extract)1500 mg Capsules (Experimental): Phaseolus Vulgaris L. is rich in alpha-amylase and alpha-glucosidase inhibitor. It has been used for calories absorption through preventing or delaying the digestion of complex carbohydrate.
  Interventions: Other: Phaseolean (White Kidney Bean Standardized Extract) 1500 mg Capsules
- Phaseolean (White Kidney Bean Standardized Extract)3000 mg Capsules (Experimental): Phaseolus Vulgaris L. is rich in alpha-amylase and alpha-glucosidase inhibitor. It has been used for calories absorption through preventing or delaying the digestion of complex carbohydrate.
  Interventions: Other: Phaseolean (White Kidney Bean Standardized Extract)3000 mg Capsules
- Placebo (Resistant Dextrin) Capsules (Placebo Comparator): Resistant dextrin is a soluble fiber, derived from wheat or corn starch and is prepared by highly controlled partial hydrolysis and repolymerization of the dextrinization process
  Interventions: Other: Placebo (Resistant Dextrin) Capsules

INTERVENTIONS:
Other: Phaseolean (White Kidney Bean Standardized Extract) 1500 mg Capsules — Mode of Usage: 2 capsules each time before 3 daily meals for consecutive 45 days.
  Route of Administration: Oral Administration with a glassful (approx. 250 mL) of water.
  Arms: Phaseolean (White Kidney Bean Standardized Extract)1500 mg Capsules
Other: Phaseolean (White Kidney Bean Standardized Extract)3000 mg Capsules — Mode of Usage: 2 capsules each time before 3 daily meals for consecutive 45 days.
  Route of Administration: Oral Administration with a glassful (approx. 250 mL) of water.
  Arms: Phaseolean (White Kidney Bean Standardized Extract)3000 mg Capsules
Other: Placebo (Resistant Dextrin) Capsules — Resistant dextrin is a soluble fiber, derived from wheat or corn starch and is prepared by highly controlled partial hydrolysis and repolymerization of the dextrinization process
  Arms: Placebo (Resistant Dextrin) Capsules

SUMMARY:
A randomized, double-blinded, placebo-controlled, single-centre, clinical safety and efficacy study in subjects with overweight or Obese Class - I, to evaluate the degree of significant weight loss by regular intake of Phaseolean (White Kidney Bean Standardized Extract).

This study is dose-response study to evaluate effectiveness of two different dosage i.e. 1500 mg Versus 3000 mg.

22 subjects will be enrolled per test treatment to complete 20 subjects per test treatment.

DETAILED DESCRIPTION:
A randomized, double-blinded, placebo-controlled, single-centre, clinical safety and efficacy study in subjects with overweight or Obese Class - I, to evaluate the degree of significant weight loss by regular intake of Phaseolean (White Kidney Bean Standardized Extract).

This study is dose-response study to evaluate effectiveness of two different dosage i.e. 1500 mg Versus 3000 mg.

22 subjects will be enrolled per test treatment to complete 20 subjects per test treatment.

The potential subjects will be screened as per the inclusion & exclusion criteria only after obtaining written informed consent from the subjects. The subjects will be instructed to visit the facility as per the below visits.

* Visit 01 (Within 30 Days): Screening, Baseline evaluations
* Visit 02 (Day 01): Enrolment & Treatment phase start
* Visit 03 (Day 21): Treatment Period, Evaluations
* Visit 04 (Day 45): Treatment Period, Evaluations & End of Study Visit
* Telephonic follow-up will be taken thrice a week (Monday, Wednesday and Friday) during an entire study to check compliance with the diet plan and study treatment.

Subjects will be pre-screened by the screening department of NovoBliss Research. Subjects will be telephonically contacted by recruiting department prior to the enrolment visit. Subjects will be instructed during screening (prior to enrolment) not to consume any weight-loss medications, or supplementation or topical anti-cellulite treatment during the study.

Eligible subjects will be randomly assigned equally to one of three groups in a 1:1:1 ratio as follows:

* Arm A (Treatment A): Subjects will be given a test treatment of 1500 mg/day (2 capsules in the morning before breakfast, 2 capsules in the afternoon before lunch and 2 capsules at night before dinner; each capsule containing 250 mg Phaseolean (White Kidney Bean Standardized Extract) along with the diet regimen and exercise as advised by the clinical nutritionist /Dietician (Diet of 2000 kcal/day throughout the study and walking exercise for 45 mins daily for consecutive 45 Days).
* Arm B (Treatment B): Subjects will be given a test treatment of 3000 mg/day (2 capsules in the morning before breakfast, 2 capsules in the afternoon before lunch and 2 capsules at night before dinner; each capsule containing 500 mg Phaseolean (White Kidney Bean Standardized Extract) along with the diet regimen and exercise as advised by the clinical nutritionist /Dietician (Diet of 2000 kcal/day throughout the study and walking exercise for 45 mins daily for consecutive 45 Days).
* Arm C (Treatment C): Subjects will be given placebo capsules (2 capsules in the morning before breakfast, 2 capsules in the afternoon before lunch and 2 capsules at night before dinner; each capsule containing 250 mg Resistant Dextrin as Placebo along with the diet regimen and exercise as advised by the clinical nutritionist /Dietician (Diet of 2000 kcal/day throughout the study and walking exercise for 45 mins daily for consecutive 45 Days).

Subjects will be followed up as per the schedule of assessments. Assessment of efficacy parameters will be done before test treatment usage on Day 1, and will be compared with after test treatments usage on Day 21 (+2 Days), & Day 45 (+2 Days) within treatments and between treatments as listed below.

* Anthropometry: Height, Weight, Body Mass Index (BMI), Hip and Waist Circumference
* Skinfold fat thickness
* Maximum Oxygen consumption (VO2)
* Vitals (Heart Rate, Blood Pressure)
* ECG and Chest X-Ray
* Blood Biochemical Parameters (Serum albumin, total protein, AST, ALT, glucose, BUN, uric acid, creatinine levels, Random Insulin)
* Biomarkers - Amylase, Lipid Profile, HbA1c
* Hedonic Questionnaires - about product perception and consumer feedback (Weight reduction, feeling of the light weight of the body, reduction of Hip and Waist circumference, reduction in skinfold fat thickness, hunger feeling, satiety level etc.)
* Digital Photographs: Body photographs with measurement of waist and hip circumference - before test treatment usage and after test treatment usage

ELIGIBILITY:
Inclusion Criteria:

The subject must fulfil all of the following inclusion criteria to be eligible for participation in the study unless otherwise specified.

1. Age: 18 to 50 years (both inclusive) at the time of consent.
2. Sex: Healthy non-pregnant/non-lactating females and Males.
3. Female of childbearing potential must have a reported negative pregnancy during screening and the end of the study.
4. Subject is generally in good health and willing to reduce weight.
5. Overweight to Obese Class - I, BMI between or equal to 25 to 35 kg/m2, or total fat percentage reaching: men > 25% and women > 30% using Karada Scan.
6. Willing to observe dietetic plan in accordance with dietitian evaluation,
7. Able and willing to participate in the study by complying with the protocol procedures.
8. Subject is willing to forgo liposuction procedures or any weight loss therapy 3 months prior to and for the duration of the study.
9. Subject is able to remain on stable doses of contraceptive or replacement hormonal therapy, including no therapy, 6 weeks prior to and for the duration of the study.
10. If the female subject is of childbearing potential, is practicing and agrees to maintain an established method of birth control (IUD, hormonal implant device/injection, regular use of birth control pills or patch, diaphragm, condoms with spermicide or sponge with spermicidal jelly, cream or foam, partner vasectomy or abstinence). Females will be considered as non-childbearing potential if they are surgically sterile, have been post-menopausal for at least 1 year or have had a tubal ligation.
11. If currently using hormonal contraception, has been using this form of contraception for at least 6 months and agrees to continue using the same contraception for the duration of the study.
12. Subject is willing to participate in exercise program (Daily, 45 mins brisk walking for consecutive 45 Days of treatment period) and recording to subject diary card.
13. Subject is willing to come in fasting state for every study visit.
14. Subject is agree to consume a vegetarian/non-vegetarian diet of approximately 2000 kcal/day (14% protein, 25%Fat and 61% carbohydrate).
15. Subject is willing to give written informed consent and are willing to follow the study procedure

Exclusion Criteria:

Subjects must not be enrolled in the study if they meet any one of the following criteria:

1. Subject has a history of allergy or sensitivity to the test treatments ingredients.
2. Subject who has a history of allergy with products containing beans, white kidney beans.
3. Subjects BMI is between less than 25 and greater than 35 kg/m2.
4. Subjects having past or present history or clinically significant findings indicating cardiovascular disease, type 2 diabetes mellitus, hypertension, endocrine, pulmonary, neurological or psychological disorders, hypo or hyperthyroidism and renal disorders.
5. Subjects having drug and alcohol abuse.
6. Smokers and tobacco users.
7. Subjects having more than 5 kg variation in body weight within 3 months before study entry.
8. Subjects using other weight loss medications, as well as stimulants, laxatives or diuretics taken solely for the purpose of weight loss.
9. Undergone surgery before 30 days of screening or planning to undergo surgery within the study period.
10. Subjects having chronic diarrhoeal disorders, cancer, hepatic dysfunction, and human immunodeficiency virus (HIV) infection.
11. Participation in other drugs, investigational medicinal product, any herbal products and/or cosmetics intended to weight loss clinical trials within 3 months before enrolment in this trial.
12. Any other diseases/co-morbidity that is considered by the Investigator as an exclusion.
13. With severe hepatic and/or renal impairment, liver enzyme level (ALT and/or AST) is greater than 2.5 times the upper normal limit.
14. Taking antibiotic therapy, anti-depressant treatment or treatment related to anxiety in the month preceding the study,
15. Taking anti-depressant treatment or treatment related to anxiety Subject in a state of depression.
16. Non-stable weight during the last 6 months (>5% change in total weight)
17. Consuming food supplements or functional foods known to have an influence on weight management in the month preceding the inclusion and/or likely to take during the test
18. Following or having followed a hypocaloric diet (energy intake <1,500 kCal/day) in the month preceding inclusion and/or likely to undertake this diet during the test.
19. Diagnosed eating disorders (bulimia, anorexia nervosa, vomiting),
20. Using topical anti-cellulite treatments
21. Pregnant or breastfeeding or planning to become pregnant during the study period.
22. Subject has a history of chronic illness which may influence the cutaneous state.
23. Subjects participating in other similar nutraceuticals, food, supplemental or therapeutic trials within the last four weeks.
24. Any other condition which could warrant exclusion from the study, as per the Investigator's discretion

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Change in Weight (Unit: Kg) | Day 1 (inclusion) to 45 Days
  Mean percentage change in Body Weight in the overweight and Obese Class - I population (Males and Females) between the treatment and placebo group
Change in BMI (Unit: Kg/m2) | Day 1 (inclusion) to 45 Days
  Mean percentage change in BMI in the overweight and Obese Class - I population (Males and Females) between the treatment and placebo group

SECONDARY OUTCOMES:
Percentage of subjects loosing weight | From baseline (i.e. Day 1) to Day 21, Day 45
  To evaluate the effectiveness of the test treatment in terms of percentage of subjects loosing weight between the treatment and placebo group
Change in Hip, Waist, and Thigh Circumference | From baseline (i.e. Day 1) to Day 21, Day 45
  To evaluate the effectiveness of the test treatment for change in Hip, waist, and thigh circumference between the treatment and placebo group
Change in total Body fat | From baseline (i.e. Day 1) to Day 21, Day 45
  To evaluate the effectiveness of the test treatment for change in total body fat by measuring skinfold fat thickness between the treatment and placebo group
Change in random blood sugar | From baseline (i.e. Day 1) to Day 21, Day 45
  To evaluate the effectiveness of the test treatment for change in random blood sugar between the treatment and placebo group
Change in HbA1C | From baseline (i.e. Day 1) to Day 45
  To evaluate the effectiveness of the test treatment for change in HbA1C between the treatment and placebo group
Change in Lipoprotein lipids (HDL, LDL, Triglyceride, and Cholesterol) | From baseline (i.e. Day 1) to Day 45
  To evaluate the effectiveness of the test treatment for change in Lipoprotein Lipids (HDL, LDL, Triglyceride, and Cholesterol) between the treatment and placebo group
Change in Serum Creatinine | From baseline (i.e. Day 1) to Day 45
  To evaluate the effectiveness of the test treatment for change in Serum Creatinine between the treatment and placebo group
Change in Serum Amylase | From baseline (i.e. Day 1) to Day 45
  To evaluate the effectiveness of the test treatment for change in Serum Amylase between the treatment and placebo group
Change in AST and ALT levels | From baseline (i.e. Day 1) to Day 45
  To evaluate the effectiveness of the test treatment for change in AST and ALT levels between the treatment and placebo group
Change in blood biochemical parameters (Serum Albumin, Total Protein, Blood Urea Nitrogen (BUN), Uric Acid, Random Insulin | From baseline (i.e. Day 1) to Day 45
  To evaluate the effectiveness of the test treatment for change in blood biochemical parameters (Serum Albumin, Total Protein, Blood Urea Nitrogen (BUN), Uric Acid, Random Insulin between the treatment and placebo group
Improvement in Maximum Oxygen Consumption (VO2) | From baseline (i.e. Day 1) to Day 45
  To evaluate the effectiveness of the test treatment for improvement in Maximum Oxygen Consumption between the treatment and placebo group
Change in BMI | From baseline (i.e. Day 1) to Day 21, Day 45
  To evaluate the effectiveness of the test treatment for change in BMI between the treatment and placebo group
Change in Heart rate | From baseline (i.e. Day 1) to Day 21, Day 45
  To evaluate the effectiveness of the test treatment for change in Heart rate between the treatment and placebo group
Change in Electrocardiogram (P wave, QRS interval, QT interval, PR interval) | From baseline (i.e. Day 1) to Day 45
  To evaluate the effectiveness of the test treatment for change in Electrocardiogram (P wave, QRS interval, QT interval, PR interval) between the treatment and placebo group
Change in Blood Pressure (Both) | From baseline (i.e. Day 1) to Day 21, Day 45
  To evaluate the effectiveness of the test treatment for change in Blood Pressure (Both) between the treatment and placebo group
Test treatment perception and consumer feedback on weight reduction, feeling of the light weight of the body, reduction of hip and waist circumference, reduction in skinfold fat thickness, hunger feeling, satiety level. | From baseline (i.e. Day 1) to Day 21, Day 45
  To evaluate the Effect of test treatment in terms of product perception and consumer feedback weight reduction, feeling of the light weight of the body, reduction of hip and waist circumference, reduction in skinfold fat thickness, hunger feeling, satiety level - using hedonic questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Dr Nayan K Patel, MBBS, Principal Investigator — Medical Director
Locations (1):
- NovoBliss Research Pvt Ltd, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No